CLINICAL TRIAL: NCT05563467
Title: A Multicentre, Open-label Phase 2 Study to Evaluate the Efficacy and Safety of Pembrolizumab in the Treatment of Advanced, Progressive Adrenocortical Carcinoma.
Brief Title: Pembrolizumab in the Treatment of Advanced, Progressive Adrenocortical Carcinoma.
Acronym: PEMBR-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Biostat Sp. z o.o. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEMBR-01
Record Dates: First submitted 2022-08-23; First posted 2022-10-03 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Adrenocortical Carcinoma
Keywords: advanced adrenocortical carcinoma; progressive adrenocortical carcinoma; pembrolizumab
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab Treatment (Experimental)
  Interventions: Drug: Pembrolizumab 25 MG/ML [Keytruda]

INTERVENTIONS:
Drug: Pembrolizumab 25 MG/ML [Keytruda] — The treatment scheme will be based on pembrolizumab administered intravenously in cycles of every 3 weeks 200 mg, with supportive treatment with steroidogenesis inhibitor (metyrapone or ketoconazole) for adrenocortical carcinoma producing cortisol.

SUMMARY:
This study is a national, multicenter, interventional, phase II clinical trial on the use of pembrolizumab in advanced adrenocortical carcinoma, with confirmed progression within 6 months, following EDP or EDP-M ( etoposide, doxorubicin, cisplatin- mitotan) chemotherapy.

Adrenocortical carcinoma is a very rare entity with poor prognosis and limited therapeutic options. Only radical surgical treatment of the early stages gives a chance for complete cure, however the risk of recurrence still remains high.

The results of clinical trials conducted outside Poland indicate a possible potential role of immunotherapy as a rescue treatment for adrenocortical carcinoma after standard therapeutic methods have been exhausted.

This study will evaluate the efficacy and tolerability of treatment with the immune checkpoint inhibitor pembrolizumab in locally advanced, non-operable or metastatic adrenocortical carcinoma after first line chemotherapy failure.

The study population will include adult patients (>18 years of age) with histopathologically confirmed adrenocortical carcinoma and confirmed progression according to RECIST 1.1 within 6 months, after first line chemotherapy with the EDP and EDP-M scheme. Patients must meet the inclusion criteria and must not meet the exclusion criteria described in the PEMBR-01 study protocol. The planned number of patients in the study is 24.

The treatment regimen will be based on Pembrolizumab administered intravenously in 3 weeks cycles at a dose of 200mg. For hormonally active tumors producing cortisol, it is hypothesized that the use of pembrolizumab in combination with effective steroidogenesis inhibition may enhance the effect of immunotherapy. In the study, metyrapone or ketoconazole will be used for this purpose.

The primary endpoint of the study will be the objective response rate to the treatment. The secondary endpoints will be progression-free survival, duration of response, overall survival, and treatment safety as well as the effect of therapy on patients' quality of life.

Concurrently, the analysis of biomarkers in tumor tissue will be carried out, including tumour infiltrating lymphocytes, expression of programmed death ligand, microsatellite instability and tumour mutation burden.

ELIGIBILITY:
Inclusion Criteria:

1. Signing the informed consent form to participate in the study
2. Age over 18 years of age
3. Histopathologically confirmed adrenocortical carcinoma
4. The general condition of the patient was assessed according to the Eastern Cooperative Oncology Group (ECOG) scale <2
5. Measurable disease according to RECIST 1.1
6. Confirmed progression according to RECIST 1.1 within the last 6 months in patients, who received at least one line chemotherapy according to the EDP or EDP-M
7. Adequate function of the marrow and internal organs:

   1. hemoglobin ≥ 9g%, neutrophils> 1500 / mm3, platelets> 100 thousand / mm3
   2. bilirubin ≤ 2 x upper limit of normal (UNL), Alat, Aspat ≤ 3 x UNL (if livermetastases are present ≤ 5 x UNL)
   3. creatinine clearance > 40 ml / min
   4. coagulation parameters: INR, PT, APTT <1.5 x UNL (exception: patients undergoing anticoagulation therapy, where INR, PT, APTT remain within the therapeutic range recommended for the patient)
8. For women of reproductive age : confirmed negative pregnancy test result, and the requirement of dual barrier contraception
9. For men of reproductive age: the requirement of dual barrier contraception

Exclusion Criteria:

1. Pre-treatment with an immune checkpoint inhibitor
2. Any cancer therapy within the last 7 days (including mitotane)
3. Persistent side effects of previous anti-cancer therapy in the> G1 stage or after surgical treatment (exception: alopecia)
4. Immunosuppressive therapy present or conducted within the last 4 weeks
5. Glucocorticoid therapy in a dose higher than the replacement dose (subject to the permitted use: inhaled or topical steroids, single administration of a steroid, e.g. in case of an allergic reaction to contrast, use of mineralocorticosteroids, steroids in the course of asthma or COPD)
6. Previous allograft marrow or organ transplant
7. Current or diagnosed in the last 2 years autoimmune disease with the exception of vitiligo, psoriasis not requiring systemic treatment, autoimmune disease of the thyroid gland
8. Active or previously documented inflammatory disease of the large intestine
9. Previous non-infectious pneumonia requiring steroid therapy
10. Hepatitis B or C
11. Active tuberculosis
12. Current active infection requiring systemic treatment
13. Symptomatic, untreated central nervous system (CNS) metastases (exception: patients with asymptomatic CNS metastases with prior surgery or radiotherapy and no history of intracranial bleeding)
14. Circulatory failure NYHA ≥3
15. Corrected QT interval> 500 ms
16. Significant coexisting disease, including neoplastic, except for basal cell carcinoma of the skin, carcinoma in situ: prostate, cervix, breast
17. Other significant comorbid disease that, in the investigator's opinion, would pose risks to the patient during therapy
18. Pregnancy or breastfeeding
19. Patients requiring dialysis
20. The patient's inability to meet the requirements specified in the study protocol
21. Vaccination with live vaccine within 3 months before starting treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the effectiveness of pembrolizumab (Keytruda) in the treatment of advanced, progressive adrenocortical carcinoma. | through study completion, an average of 4 years
  Outcome will be assessed based on i.a. objective response rate (ORR).

SECONDARY OUTCOMES:
Assessment of the safety of pembrolizumab (Keytruda) in the treatment of advanced, progressive adrenocortical carcinoma. | through study completion, an average of 4 years
  Number of Adverse Events and Serious Adverse Events (AE and SAE) related and not related to treatment according to CTCAE.
Assessment of the impact of therapy on the patient's quality of life. | through study completion, an average of 4 years
  Quality of life assessed based on the QLQ-C30 questionnaire in which patients will respond during the clinical trial.

CONTACTS AND LOCATIONS:
Locations (4):
- Poland (4):
  - Maria Sklodowska-Curie National Research Institute of Oncology, Gliwice, Silesian Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki W Krakowie, Krakow
  - Uniwersytecki Szpital Kliniczny W Poznaniu, Poznan
  - Medical University Of Warsaw, Warsaw

IPD SHARING:
Plan to Share IPD: No